CLINICAL TRIAL: NCT06054945
Title: Clinical Impact of IPACK Block Addition to Suprainguinal Fascia Iliaca Block in Knee Arthroplasty Patients Under Spinal Anesthesia: A Retrospective Cohort Study
Brief Title: Clinical Impact of IPACK Block Addition to Suprainguinal Fascia Iliaca Block
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SIFIB+IPACK
Record Dates: First submitted 2023-09-15; First posted 2023-09-26 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Analgesia; Pain Management; Acute Pain
Keywords: analgesia; IPACK; SIFIB
MeSH Terms: conditions — Agnosia; Acute Pain | interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SIFIB: Patients who underwent SIFIB in knee arthroplasty patients under spinal anesthesia will be evaluated retrospectively in terms of opioid consumption and NRS scores.
  Interventions: Procedure: SIFIB (suprainguinal fascia iliaca block); Device: Patient controlled anagesia device
- SIFIB+IPACK: Patients who underwent SIFIB+IPACK blocks in knee arthroplasty patients under spinal anesthesia will be evaluated retrospectively in terms of opioid consumption and NRS scores.
  Interventions: Procedure: SIFIB (suprainguinal fascia iliaca block); Other: IPACK (Interspace between the popliteal artery and capsule of the posterior knee ); Device: Patient controlled anagesia device

INTERVENTIONS:
Procedure: SIFIB (suprainguinal fascia iliaca block) — Ultrasound guided Suprainguinal Fascia Iliaca Block for Knee Arthroplasty Patients
Other: IPACK (Interspace between the popliteal artery and capsule of the posterior knee ) — Ultrasound guided IPACK (Interspace between the popliteal artery and capsule of the posterior knee ) Block for Knee Arthroplasty Patients
  Groups: SIFIB+IPACK
Device: Patient controlled anagesia device — Those who were administered opioids with PCA as rescue analgesic in the postoperative analgesia plan on the selected dates will be included in the study.
  Other Names: PCA

SUMMARY:
In our clinic, routine suprainguinal fascia iliaca block (SIFIB) has been administered for postoperative analgesia in patients undergoing knee arthroplasty. Recently, we have introduced the IPACK (Infiltration between the Popliteal Artery and Capsule of the Knee) block to this regimen, and the aim of this retrospective study is to determine whether the addition of the IPACK block enhances the quality of analgesia.

Knee arthroplasty, also known as knee joint replacement surgery, is a common procedure performed to alleviate pain and improve joint function in patients with knee osteoarthritis or other knee-related conditions. Postoperative pain management is crucial for patient comfort and overall recovery.

In this study, we aimed to compare the two techniques mentioned earlier, namely the SIFIB (Suprainguinal Fascia Iliaca Block) and the SIFIB+IPACK, by examining the data of patients who underwent knee arthroplasty under spinal anesthesia at our clinic between January 1, 2023, and September 1, 2023.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the following criteria and whose postoperative follow-up forms were completed in full were included in the study
* Patients underwent total knee arthroplasty (TKA)
* ASA class I to III.
* operated under spinal anesthesia
* patient controlled analjgesia device was used for analgesia

Exclusion Criteria:

Patients whose data were inaccessible or had incomplete follow-up forms were excluded from the study to ensure the accuracy and reliability of our analysis.

* PCA device problems in follow up in 24 hours
* anesthesia plans were converted to general anesthesia
* spinal anesthesia failure
* peripheral blocks used other than protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: data of patients underwent total knee arthroplasty under spinal anesthesia between 01.01.2023 and 01.09.2023
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2023-09-03 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours
  Opioid consumption via PCA device

SECONDARY OUTCOMES:
NRS scores | 24 hours
  NRS scores in different time frames. In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Kusderci, M.D., Principal Investigator — Samsun University
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)